CLINICAL TRIAL: NCT06954935
Title: Effectiveness of Periorbital Massage in the Management of Nausea and Vomiting After Laparoscopic Cholecystectomy
Brief Title: Periorbital Massage for Nausea and Vomiting After Laparoscopic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Cagla Toprak, Dr, Atlas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23.12.2024 10/3
Record Dates: First submitted 2025-04-23; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Nausea; Vomiting; Laparoscopic Cholecystectomy
Keywords: nausea; voming; periorbital massage
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- periorbital massage (Experimental): The severity of nausea and frequency of vomiting of patients will be analyzed at the 2nd, 4th, 6th, 8th, 12th and 24th hours after surgery. 15 minutes before these evaluations, an electronic eye massager (irest manufacturing company, China) will be applied to the patient's eyeball (according to the manufacturer's instructions) for 15 minutes. 15 minutes after the intervention, the severity of nausea and vomiting of patients will be evaluated using the nausea numerical scale and the vomiting incidence evaluation form.
  Interventions: Other: periorbital massage
- control (No Intervention): The severity of nausea and frequency of vomiting of patients will be analyzed at 2, 4, 6, 8, 12 and 24 hours after surgery. Data collection intervals will be the same in both control and intervention groups.

INTERVENTIONS:
Other: periorbital massage — An electronic eye massager (irest manufacturing company, China) will be applied. The massager has a vibration function and massages with a warm air bag.
  Arms: periorbital massage

SUMMARY:
Laparoscopic cholecystectomy is one of the commonly used surgical treatment methods for gallbladder diseases. However, many patients experience significant nausea and vomiting after laparoscopic cholecystectomy. It is observed that approximately 20% to 30% of patients experience postoperative nausea and vomiting as the most common complaint after laparoscopic cholecystectomy. This study aims to investigate the effectiveness of periorbital massage in postoperative nausea and vomiting in patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
This study aimed to investigate the effectiveness of periorbital massage in postoperative nausea and vomiting in patients undergoing laparoscopic cholecystectomy. One group received periorbital massage, while the other group did not receive massage.

ELIGIBILITY:
Inclusion Criteria:

Those who have laparoscopic cholecystectomy surgery under general anesthesia,

* Those between the ages of 18-70,
* Those who do not have a psychiatric disease,
* Those who understand what they read and volunteer patients,
* Those who do not have a hearing or speech problem,

Exclusion Criteria:

* Patients undergoing emergency surgery,

  * Patients with psychiatric disorders
  * Patients who have taken another antiemetic drug within 24 hours before surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2025-08-25 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Apfel risk score | It will be filled half an hour before you go down for surgery.
  : Apfel Risk Score is a simple scoring used to determine the risk status of patients for PONV. Apfel Risk Score questions four factors such as being female, not smoking, having a history of PONV/motion sickness and using postoperative opioids. Each factor is evaluated as 1 point. Apfel risk score varies between 0-4 and is classified as low, medium and high risk. Apfel Risk score 0-1 is evaluated as low risk, 2 as medium risk and 3-4 as high risk.
Numerical Scale of Nausea | 0, 2, 6, 12 and 24 hours after surgery
  The numerical scale of nausea is a scale that starts with "0 (no nausea)" and ends with "10 (very severe nausea)" and is given a numerical value with 1 cm intervals. The numerical scale is one-dimensional and is mainly used to evaluate the severity of pain.
Postoperative Nausea and Vomiting Impact Scale | 0, 2, 6, 12 and 24 hours after surgery
  There are four options in the two-question scale, each with 0, 1, 2, or 3 points. The first question asks whether there is vomiting or retching, if any, and the frequency; the answers are "0" no, "1" once, "2" twice, "3" three times or more, with four options. The second question asks whether there is nausea (feeling of discomfort in the stomach and feeling like vomiting), if any, whether the feeling of nausea affects your ability to get out of bed, move around comfortably in bed, walk normally, or your daily life activities such as eating and drinking; the answers are "0" not very often, "1" sometimes, "2" often or often, and "3" always, with four options. The numerical values of the answers given to the first and second questions are added up and the result is found.

CONTACTS AND LOCATIONS:
Locations (1):
- Tuğba Albayram, Gaziantep, Turkey (Türkiye)